

## STUDY PROTOCOL

(July 30th 2019)

# Effectivity of Liquid Nutritional Supplementation in Improving Nutritional Status of Hospitalized Malnutrition Patients: A Single-Blind Randomized Controlled Trial

PRINCIPAL INVESTIGATOR: Prof. dr. Marcellus Simadibrata, PhD., SpPD-KGEH

CO-INVESTIGATOR : Prof. Dr. dr. Murdani Abdullah, SpPD-KGEH

dr. Amanda Pitarini Utari, SpPD-KGEH

dr. Virly Nanda Muzellina, SpPD

Faculty of Medicine
Universitas Indonesia
(FMUI)

## Title

Effectivity of Liquid Nutritional Supplementation in Improving Nutritional Status of Hospitalized Malnutrition Patients: A Single-Blind Randomized Controlled Trial

### Background

Malnutrition is a common problem that is found in hospitalized patients. A study by Allard et al<sup>1</sup> found that in Canada, 45% of hospitalized patients had malnutrition. Another studies in Europe, 20-30% of hospitalized patients also had malnutrition.<sup>2,3</sup> Lim et al<sup>4</sup> also conducted a study and found malnutrition in 27-39% subjects who were hospitalized. Malnutrition is a condition which there were unbalanced energy, protein or other nutrition that results in underweight or overweight. Malnutrition in hospitalized patients is due to unfullfiled nutrient intake, malabsorption, nutrient loss due to main disease or increased metabolic demand.<sup>5,6</sup>

Recent studies showed that malnutrition increases morbidity and mortality. Malnutrition also extends hospitalisation duration and recovery time. These will increase hospitalisation cost. <sup>7-9</sup> Therefore, nutrition is an important key in malnutrition treatment. Nutritional supplementation can be given in improving nutritional status. Liquid form is a alternative in supplying nutrition to hospitalized patients since the consistency made it easier to swallow. Nowadays nutritional supplement in liquid form is available from commercial product or hospital product. Therefore, we need a study to know effectivity liquid nutritional supplement from hospital product in malnutrition hospitalized patients.

## **Objective**

#### General objective

To know the effectivity of liquid nutritional supplementation in malnutrition hospitalized patients

#### Specific objectives

- 1. To know the change of Body Mass Index (BMI) post liquid nutritional supplementation
- 2. To know the change of Subjective Global Assessment (SGA) rank post liquid nutritional supplementation
- 3. To know the change of hemoglobin level post liquid nutritional supplementation
- 4. To know the change of prealbumin level post liquid nutritional supplementation

- 5. To know the change of Blood Urea Nitrogen (BUN) level post liquid nutritional supplementation
- 6. To know the change of lipid profile level post liquid nutritional supplementation
- 7. To know the change of blood glucose level post liquid nutritional supplementation
- 8. To know the change of body fat percentage post liquid nutritional supplementation
- 9. To know the change of handgrip strength test score post liquid nutritional supplementation

#### Methods

## Study Design

This research is a single blind, randomized clinical trial method. Analysis will be conducted pre and post administration: control (standard liquid nutritional supplement as placebo), intervention (liquid nutritional supplement from hospital product) 2 times daily for 14 days.

## Location and Time

This research will be conducted on Indonesia from August 2019 to December 2020

## Population and Subject

#### **Population**

The population of this research is hospitalized patients with malnutrition in Indonesia

#### Subjects Criteria

- Inclusion criteria
  - 1. Subjects aged  $\geq$  18 years old to 60 years old
  - Malnutrition hospitalized patient based on European Society for Clinical Nutrition and Metabolism (ESPEN) 2015 criteria
  - 3. Agreed to participate

#### - Exclusion criteria

- 1. Malignancy
- 2. Chronic kidney disease stage III-V
- 3. Decompensated hepatic cirrhosis
- 4. Allergic to milk or lactose intolerance
- 5. Could not be randomised and participate in this study by clinical judgement

## Drop Out Criteria

Drop out subjects are subjects who have signed the informed consent but decide to withdraw before research is completed

# Estimated Sample Size

Minimum sample size is determined using the following equation for proportion equation.

N1 = N2 = 
$$\frac{(Z_{\alpha}\sqrt{2PQ} + Z_{\beta}\sqrt{P_1Q_1 + P_2Q_2})^2}{(P_1 - P_2)^2}$$

Description:

$$Z\alpha = 1.96$$
  $Z\beta = 0.84$ 

$$P_1 - P_2 = 0.2$$
  $P_1 = 0.15^{10}$ 

N1 = N2 = 62.41, thus with predicted drop out 10% the minimal sample for each group is 69 subjects

#### Randomization

Randomization is generated by computer and subjects will be given code and divided into two groups (control and intervention). Only researchers are blinded to treatment. Subjects can't be blinded since the taste between intervention and placebo is obvious.

#### <u>Variables</u>

#### Independent Variables

- 1. Intervention: administration of liquid nutritional supplement from hospital product 2 times daily
- 2. Control (placebo): administration of standard nutritional product 2 times daily

## **Dependent Variables**

- 1. Body Mass Index (BMI)
- 2. Hemoglobin, prealbumin, Blood Urea Nitrogen (BUN), lipid profile, blood glucose from blood samples
- 3. Subjective Global Assessment (SGA) rank
- 4. Body fat percentage from Bioelectrical Impedance Analysis (BIA)
- 5. Handgrip strength score from handgrip strength test

#### **Procedure**

1. Eligibility assessment

The subjects will be assessed for eligibility using inclusion and exclusion criteria.

- 2. Subjects sign the informed consent form
- 3. Randomization
- 4. Pre-administration
- 6. Before administration of liquid nutritional supplement either from commercial or hospital product or placebo based on randomization, subjects will be analysed for his/her BMI, hemoglobin, prealbumin, Blood Urea Nitrogen (BUN), lipid profile, blood glucose, Subjective Global Assessment (SGA) rank, body fat percentage and handgrip strength score. Subject will also be examined for his/her skinfold and mid upper arm circumference.
- Administration (14 days)
   Subjects will be given liquid nutritional supplement and placebo that will be taken two times daily for 14 days.
- 6. Compliance monitoring

Compliance monitoring of administration is conducted by the investigators coordinating with his/her family, nurses and doctors in the hospital while patient is hospitalized

7. Post administration

After 14 days, the subjects will be analysed for his/her BMI, hemoglobin, prealbumin, Blood Urea Nitrogen (BUN), lipid profile, blood glucose, Subjective Global Assessment (SGA) rank, body fat percentage and handgrip strength score.

- 8. Data analysis
  - a. Normality analysis using Kolmogorov-Smirnov (Normally distributed if p>0.05)
  - b. Bivariate analysis by comparing numeric data between two groups: if data is normality distributed using T-test, if not using Mann-Whitney test (significant if p<0.05)
  - c. Bivariate analysis by comparing categorical data between two groups: if data is normality distributed using T-test, if not using Mann-Whitney test (significant if p<0.05)
  - d. Bivariate analysis by comparing numeric data between preadministration and postadministration: if data is normality distributed using paired T-test, if not using Wilcoxon test (significant if p<0.05)

e. Bivariate analysis by comparing categorical data between preadministration and postadministration: if data is normality distributed using Mc Nemar test, if not using Wilcoxon test (significant if p<0.05)

## Study flow chart



Day 0: BMI, hemoglobin, prealbumin, Blood Urea Nitrogen (BUN), lipid profile, blood glucose, Subjective Global Assessment (SGA) rank, body fat percentage and handgrip strength score assessment



Day 14: BMI, hemoglobin, prealbumin, Blood Urea Nitrogen (BUN), lipid profile, blood glucose, Subjective Global Assessment (SGA) score, body fat percentage and handgrip strength score assessment

#### Ethical committee approval

Approval from the Ethical Committee at the Faculty of Medicine Universitas Indonesia must be obtained before starting the trial.

#### References

1. Allard JP, Keller H, Jeejeebhoy KN, et al. Malnutrition at Hospital Admission - Contributors and Effect on Length of Stay: A Prospective Cohort Study From the Canadian Malnutrition Task

- Force. J Parenter Enter Nutr. 2015;40(4):487-497.
- 2. Schindler K, Pernicka E, Laviano A, et al. How nutritional risk is assessed and managed in European hospitals: A survey of 21,007 patients findings from the 2007-2008 cross-sectional nutritionDay survey. Clin Nutr. 2010;29(5):552-559.
- 3. Álvarez-Hernández J, Planas Vila M, León-Sanz M, et al. Prevalence and costs of malnutrition in hospitalized patients; the PREDyCES Study. Nutr Hosp. 2012;27(4):1049-1059.
- 4. Lim SL, Ong KCB, Chan YH, Loke WC, Ferguson M, Daniels L. Malnutrition and its impact on cost of hospitalization, length of stay, readmission and 3-year mortality. Clin Nutr. 2012;31(3):345-350.
- 5. Meijers JMM, van Bokhorst-de van der Schueren MAE, Schols JMGA, Soeters PB, Halfens RJG. Defining malnutrition: Mission or mission impossible? *Nutrition*. 2010;26(4):432-440.
- 6. Correia MITD, Perman MI, Waitzberg DL. Hospital malnutrition in Latin America: A systematic review. *Clin Nutr*. 2016;36(4):958-967.
- 7. Ray S, Laur C, Golubic R. Malnutrition in healthcare institutions: A review of the prevalence of under-nutrition in hospitals and care homes since 1994 in England. *Clin Nutr.* 2013;33(5):829-835.
- 8. Rahman A, Wu T, Bricknell R, Muqtadir Z, Armstrong D. Malnutrition Matters in Canadian Hospitalized Patients: Malnutrition Risk in Hospitalized Patients in a Tertiary Care Center Using the Malnutrition Universal Screening Tool. *Nutr Clin Pract*. 2015;30(5):709-713.
- 9. Khalatbari-Soltani S, Marques-Vidal P. The economic cost of hospital malnutrition in Europe; a narrative review. *Clin Nutr ESPEN*. 2015;10(3):e89-e94.
- 10. Esmarie van Tonder, Lynn Gardner, Saskia Cressey, Reinette Tydeman-Edwards & Karin Gerber. Adult malnutrition: prevalence and use of nutrition-related quality indicators in South African public-sector hospitals, South African Journal of Clinical Nutrition 2019;32(1):1-7.